CLINICAL TRIAL: NCT01004588
Title: The Effects of Resistance Type Exercise Training and Protein Supplementation on Skeletal Muscle Mass, Strength, and Muscle Characteristics in Healthy Elderly Men and Women
Brief Title: The Effects of Resistance Training and Protein Supplementation in Healthy Elderly Men and Women.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Top Institute Food and Nutrition (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MEC 09-3-056
Record Dates: First submitted 2009-10-26; First posted 2009-10-30 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: Muscle Loss in Elderly
Keywords: elderly; sarcopenia; protein drink; resistance training
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Protein drink (Experimental): protein drink
  Interventions: Dietary Supplement: Protein drink
- Placebo drink (Placebo Comparator): Placebo drink
  Interventions: Dietary Supplement: placebo drink

INTERVENTIONS:
Dietary Supplement: Protein drink — total of 15 g protein/d in a protein drink consumed every morning after breakfast during 24 weeks
  Arms: Protein drink
Dietary Supplement: placebo drink — subjects consume a placebo drink every morning after breakfast over a period of 24 weeks.
  Arms: Placebo drink

SUMMARY:
The main objective of this study is to examine the effects of resistance type exercise training combined with nutritional support on body composition and muscle characteristics in healthy elderly men and women. For a comprehensive insight into the potential underlying mechanisms of the intervention effects on whole body-, muscle- and myocellular level, a broad range of tests will be performed before, during, and after the intervention period.

ELIGIBILITY:
Inclusion Criteria:

* over 65 years
* healthy men and women

Exclusion Criteria:

* cardiovascular disease
* COPD
* Parkinson
* rheumatoid arthritis
* musculoskeletal/orthopaedic disorders
* cognitive impairment
* subjects with metal implants

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-11; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Change in muscle mass measured by DXA-scan and CT-scan | 0, 12 and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Marika Leenders, MSc, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University, Maastricht, Netherlands